CLINICAL TRIAL: NCT05885087
Title: 'Extended Balloon Catheter' Labour Induction; a Single Arm Pilot Trial
Brief Title: 'Extended Balloon Catheter' Labour Induction; a Single Arm Pilot Trial'
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Botswana (Other)
Responsible Party: Principal Investigator, Lorato Matshitsa, Senior Resident, Department of Obstetrics and Gynecology, University of Botswana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UBR/RES/IRB/BIO/GRAD/145
Record Dates: First submitted 2023-05-07; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Labor, Induced
Keywords: foley/balloon catheter; labor induction; favorable cervix

STUDY DESIGN:
Intervention Model Description: single group prospective trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Foley/Balloon catheter arm (Experimental): Participants were assessed as having a favourable cervix using the modified Bishop score of equal to or more than 7. Three Foley balloon catheters attached side by side were inflated with 60mls each and a gentle traction of 250mls water applied.
  Interventions: Device: Foley or balloon catheter

INTERVENTIONS:
Device: Foley or balloon catheter — Three Foley balloon catheters attached side by side were inflated with 60mls each and a gentle traction of 250mls water applied.

SUMMARY:
The overall aim of the single arm pilot study was to assess the effectiveness, safety and acceptance of the 'extended balloon catheter' as a method of induction of labour in women receiving care at Princess Marina Hospital(PMH) in Gaborone, Botswana.

The main questions it aimed to answer were whether 'extended balloon catheter' is an effective method of labour induction, whether it results in increased adverse events for the mother and baby and whether it is associated with increased mother satisfaction.

Participants were assessed as having a favourable cervix using the modified Bishop score of equal to or more than 7. Three Foley balloon catheters attached side by side were inflated with 60mls each and a gentle traction of 250mls water applied. Delivery interval (time of induction to time of delivery), mode of delivery and Apgar scores were recorded. Adverse maternal and neonatal outcomes were recorded. Participants' satisfaction with the method of induction was assessed using a descriptive scale.

DETAILED DESCRIPTION:
Labour induction is indicated when the benefits to the mother and/or foetus of discontinuing the pregnancy outweigh the risks of awaiting spontaneous onset of labour. However, induction of labour is not without risk and the World Health Organisation recommends induction of labour be performed with a clear medical indication and when the expected benefits outweigh potential harms. Established indications for induction of labour include gestational age of 41 completed weeks or more, prelabour rupture of amniotic membranes, hypertensive disorders, maternal medical complications, foetal growth restriction, chorioamnionitis, multiple pregnancy, vaginal bleeding and other complications.

The ideal method for induction should be safe for both the mother and baby, cost effective and not require extensive monitoring. Trans-cervical extra-amniotic Foley catheter placement has been shown to be the safest method of labour induction with fewer maternal and neonatal side effects such as uterine hyperstimulation and changes in foetal heart rate during labour than prostaglandins or oxytocin. It has also been shown that there were no significant differences between caesarean and vaginal deliveries between Foley catheter, prostaglandins and oxytocin, although labour was shown to last longer after induction with Foley catheter than with prostaglandins and oxytocin. These factors can therefore potentially influence the women's preference for either method.

Foley catheter has generally been used for labour induction with an unfavourable cervix and once the cervix is favourable or the Foley method is unsuccessful, prostaglandins or oxytocin with amniotomy are used. In lower and middle income countries like Botswana where patient monitoring during induction of labour and labour is limited and mostly intermittent, mainly due to the limited or lack of monitoring devices to detect uterine hyperstimulation or foetal heart rate changes, a high patient to midwife ratio, and a high HIV prevalence, it may be preferable to avoid amniotomy and risks associated with hyperstimulation with exogenous oxytocin or prostaglandins. There are no randomized trials of Foley catheter induction with a favourable cervix reported in the Cochrane review of mechanical methods of labour induction. To optimize the likelihood of delivery without recourse to amniotomy and oxytocin or prostaglandins, 'extended balloon catheter' has been proposed as a method of continuing induction and augmentation with a Foley catheter rather than switching to other methods.

The purpose of this proposed single arm pilot trial was to test this novel idea of using 'extended balloon catheter' for induction of labour in women with favourable cervix in Botswana, and assess its effectiveness, safety to both the mother and baby as well as patient satisfaction with the procedure. Findings from this study will guide clinical protocols on how to utilize the safest available option for optimal maternal and neonatal outcomes as well as offer options and evidence for counselling women for whom prostaglandins or oxytocin are contraindicated or for use with caution in Botswana and elsewhere.

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years or older without serious morbidity due for labour induction, who give consent to participate.
* Cervix considered too far dilated to retain a single balloon, or single balloon has fallen out while not yet in labour.
* Bishop score of equal or more than 7.
* Nulliparous and multiparous
* Singleton and cephalic
* Gestation >37+0 weeks
* Estimated fetal weight <4kg

Exclusion Criteria:

* Previous caesarean delivery
* Very urgent labour induction indications (eg eclampsia, preeclampsia with severe features)
* Ruptured membranes

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Successful labor induction | Enrolment until 60 hours
  Successful labor induction defined as vaginal birth within 60 hours.

SECONDARY OUTCOMES:
Adverse event | Enrolment until discharge from hospital, or up to 2 weeks
  Any adverse maternal and fetal outcomes in participants
Acceptability | Enrolment until discharge from hospital, or up to 2 weeks
  Satisfaction with the procedure as defined by postpartum questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: JUSTUS HOFMEYR, DSc, Study Director — University of Botswana
Locations (1):
- Princess Marina Hospital, Gaborone, South-East District, Botswana

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, consent form and data collection tool.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: within 5 years after study completion.
Access Criteria: reasonable request in the context of an approved protocol